CLINICAL TRIAL: NCT00235911
Title: Effects of Symbicort Single Inhaler Therapy on Bronchial Hyper Responsiveness, Asthma Control and Safety in Mild to Moderate Asthmatics in General Practice, Compared to Usual Care Therapy
Brief Title: Symbicort Single Inhaler Therapy for Asthma in a General Practice Setting
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BN-00S-0011
Record Dates: First submitted 2005-10-07; First posted 2005-10-12 (Estimated); Last update posted 2011-01-24 (Estimated); Status verified 2011-01

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Budesonide

INTERVENTIONS:
Drug: budesonide/formoterol Turbuhaler

SUMMARY:
The primary objective is to compare the effects of Symbicort SiT and treatment according to NHG-guidelines on bronchial hyperresponsiveness in asthmatic patients, as measured by PD20 histamine, and to validate the Bronchial Hyperresponsiveness Questionnaire (BHQ).

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of mild to moderate asthma, FEV1 ³ 60% of predicted normal values pre-bronchodilator, daily use of inhaled GCS during the last 3 months

Exclusion Criteria:

* Regular need of >4 inhalations of a short-acting b2-agonist/day, known or suspected hypersensitivity to any of the investigational drugs or inhaled lactose, use of any b-blocking agent, having smoked ³10 pack-years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100
Dates: Start 2003-09; Primary Completion 2006-10 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Change in PD20 histamine

SECONDARY OUTCOMES:
number of asthma-control days, time to first mild asthma exacerbation, number of mild asthma exacerbation days, asthma symptom scores (day and night), FEV1, PEF (morning and evening), Number of inhalations with iGCS and mean dose of iGCS

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca Netherlands Medical Director, MD, Study Director — AstraZeneca
Locations (2):
- Netherlands (2):
  - Research Site, Appingedam
  - Research Site, Groningen

REFERENCES:
- [Derived] Riemersma RA, Postma D, van der Molen T. Budesonide/formoterol maintenance and reliever therapy in primary care asthma management: effects on bronchial hyperresponsiveness and asthma control. Prim Care Respir J. 2012 Mar;21(1):50-6. doi: 10.4104/pcrj.2011.00090. PMID 22015542